CLINICAL TRIAL: NCT03095131
Title: Assessment of the Clinical Efficacy of the Heart Spectrum Blood Pressure Monitor for Diagnosis of Atrial Fibrillation: An Unblinded Clinical Trial
Brief Title: Assessment of the Clinical Efficacy of the Heart Spectrum Blood Pressure Monitor for Diagnosis of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostar Meditech Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TMU JIRB No.: N201510061
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation
Keywords: Heart Spectrum Blood Pressure MonitorHeart Spectrum
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 12-lead ECG (Experimental)
  Interventions: Device: Heart Spectrum Blood Pressure Monitor

INTERVENTIONS:
Device: Heart Spectrum Blood Pressure Monitor — The Heart Spectrum Blood Pressure Monitor provides a convenient and effective filtering application compared with traditional methods that require a visit to a physician for a 12-lead ECG.

SUMMARY:
Question: Is 12-lead electrocardiography (ECG) the most accurate and convenient diagnostic method for atrial fibrillation (AF)? Findings: The Heart Spectrum Blood Pressure Monitor can be used at home, and is capable of determining the occurrence of AF. Three measurement methods were used in this study. The sensitivity, specificity, PPV, and NPV of the methods used are between 90% and 100%, and the Heart Spectrum Blood Pressure Monitor can be effectively applied to AF detection.

Meaning: The Heart Spectrum Blood Pressure Monitor can be used at home and can replace the need for an in-office ECG, thereby accomplishing meaningful telecare.

DETAILED DESCRIPTION:
Importance: Atrial fibrillation (AF) is the most common arrhythmia. The most common diagnostic method, 12-lead ECG, can record episodes of arrhythmia from which the type and severity can be determined. The Heart Spectrum Blood Pressure Monitor (P2, OSTAR Meditech Corp.) is used to measure cardiovascular pressure change, with fast Fourier transform (FFT) analysis, to obtain the heart rate frequency variability and accurate blood pressure data.

Objective: To compare the diagnostic efficacy of the Heart Spectrum Blood Pressure Monitor with a 12-lead ECG in patients with AF. Three measurement methods were used in this study: blood pressure, mean arterial pressure (MAP) which is calculated from individual blood pressure as constant pressure, and a constant pressure 60 mmHg, in order to analyze the heart index and compare it with simultaneous 12-lead ECG.

Design: The physician used a 12-lead ECG and the Heart Spectrum Blood Pressure Monitor simultaneously. The Heart Spectrum Blood Pressure Monitor used an FFT analysis for the diagnosis of AF; the findings were compared with the readings from the 12-lead ECG.

Setting: This unblinded clinical trial was conducted at the Emergency Room of Taipei Medical University Hospital.

Participants: Twenty-nine subjects with AF and 33 without AF, aged 25 to 97 years (mean: 63.5 years), were included.

Intervention(s) for clinical trials Subjects who had been exposed to high frequency surgical equipment during testing, those with cardiac pacemakers or implantable defibrillators, and pregnant women were excluded.

Trial Registration: TMU JIRB No.: N201510061

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 20 years of age who had been diagnosed with AF using 12-lead ECG, or were healthy (without AF) were included.

Exclusion Criteria:

* Subjects who had been exposed to high frequency surgical equipment during testing, those with cardiac pacemakers or implantable defibrillators, and pregnant women were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
The Heart Spectrum Blood Pressure Monitor used an FFT analysis for the diagnosis of AF; the findings were compared with the readings from the 12-lead ECG. | monitoring for about 60 seconds per test
  In the emergency room, when medical staff found patients with AF, they informed the research physicians to study the case. The Heart Spectrum Blood Pressure Monitor was compared with 12-lead ECG (ELI 250) after written informed consent was obtained from the patient. The results were interpreted by the emergency physician. Finally, the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) were analyzed to evaluate the clinical efficacy.

IPD SHARING:
Plan to Share IPD: No